CLINICAL TRIAL: NCT00821002
Title: An Open-Label, Phase 2 Study of Punctal Placement of the Latanoprost Punctal Plug System (L-PPDS) in Subjects With Ocular Hypertension (OH) or Open-Angle Glaucoma (OAG)
Brief Title: A Phase 2 Study of Punctal Placement of the Latanoprost Punctal Plug Delivery System (L-PPDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Collaborators: QLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPL GLAU 05
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plug placement (Experimental)
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: Latanoprost — Comparison of punctal plug placement between upper and lower puncta

SUMMARY:
The study objective is to compare IOP and safety outcomes based on plug placement (upper or lower puncta).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Diagnosed with bilateral Open-Angle Glaucoma or Ocular Hypertension

Exclusion Criteria:

* Uncontrolled medical conditions
* Subjects who wear contact lenses
* Subjects requiring chronic topical artificial tears, lubricants, and /or requiring any other chronic topical medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure change from baseline (mmHg) | 6 weeks

SECONDARY OUTCOMES:
Number of subjects with adverse events | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Cuzanni, MD, MSc, Study Director — QLT Inc.
Locations (1):
- Menlo Park, California, United States